CLINICAL TRIAL: NCT06368765
Title: Effects of Oral Rehydration Solution on Dehydration Recovery in Adults
Brief Title: Oral Rehydration Solution and Dehydration Recovery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in Research Focus
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: BL72
Record Dates: First submitted 2024-04-12; First posted 2024-04-16 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration | interventions — World Health Organization oral rehydration solution; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Rehydration Solution (Experimental): Oral rehydration solution with carbohydrate
  Interventions: Other: Oral Rehydration Solution (ORS)
- Water (Experimental): Water with flavor
  Interventions: Other: Water

INTERVENTIONS:
Other: Oral Rehydration Solution (ORS) — Participants will be administered the ORS during one of the study visits
  Arms: Oral Rehydration Solution
Other: Water — Participants will be administered water during one of the study visits
  Arms: Water

SUMMARY:
This is a prospective, randomized, controlled, blinded, crossover, study to evaluate the effects of an oral hydration solution.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18 to 40 years of age.
* Participant has a body mass index (BMI) ≥ 18 and ≤ 30 kg/m2
* Participant reports having a moderate to heavy sweat rate when physically exerted or in extreme heat.
* Participant is male or non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
* Participant has a systolic blood pressure of < 130 mm Hg and a diastolic blood pressure < 90 mm Hg, without the use of anti-hypertensive medications.
* Participant reports no predisposing cardiovascular conditions.
* If female, participant has a regular menstrual cycle.
* Participant is willing to consume grape-flavored beverages during the study.
* If participant is on chronic medication, the dosage must be constant for at least 2 months prior to first study visit and able to maintain medication type and dose throughout duration of study.
* Participant is weight-stable for the two months prior to screening visit
* Participant has voluntarily signed and dated an informed consent form (ICF), approved by an IRB, and provided applicable privacy regulation authorization prior to any participation in the study.
* Participant has no known intolerance or allergy to ingredients in study products.
* Participant is willing to refrain from using saunas or hot tubs for the duration of the study.
* Participant is able and willing to follow study procedures and complete any forms or assessments needed during the study.

Exclusion Criteria:

* Participant is a current, and including the past 8 weeks, participant in a weight-conscious sport such as but not limited to wrestling, powerlifting, boxing, rowing, gymnastics or any martial arts, with participation defined as ≥ 3x weekly training.
* Participant is currently, and for the past 4 weeks or longer: running >40 miles per week on average, cycling >80 miles per week on average or swimming >20,000 yards per week on average.
* Participant is participating in another study that has not been approved as a concomitant study
* Participant has used a sauna in the past 4 weeks.
* Participant uses any form of tobacco or nicotine, or other controlled substance not prescribed by a physician.
* Participant has previous history with heat illness or injury that resulted in a visit to a medical center in the past 12 months.
* Participant has an eating disorder, severe dementia or delirium, history of significant neurological or psychiatric disorder, alcoholism, substance abuse or other conditions that may interfere with study product consumption or compliance with study protocol procedures.
* Participant is currently taking or has taken antibiotics within 6 weeks of enrollment.
* Participant is currently taking or has taken a diuretic within 1 week of enrollment.
* Participant has been diagnosed with the following according to self-report:

  * Recent or current acute or chronic infections including but not restricted to respiratory infections, diarrhea, Hepatitis B or C, HIV infection or tuberculosis
  * Severe gastrointestinal disorders such as celiac disease, short bowel syndrome, pancreatic insufficiency, or cystic fibrosis
  * Metabolic [including diabetes], renal, hepatic, or respiratory disease
  * Active malignancy
  * Polycystic ovary disease
  * Any other clinically significant medical condition, which in the investigator's opinion, makes him or her unsuitable for inclusion in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2024-07-08 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Plasma Volume | Through Study completion, an average of 2 weeks
  Calculated Change in Plasma Volume

SECONDARY OUTCOMES:
Body Mass | Through Study completion, an average of 2 weeks
  Change in Body Mass
Hydration Status Urine | Through Study completion, an average of 2 weeks
  Change in Urine Osmolality
Blood Biomarker - Plasma Osmolality | Through Study completion, an average of 2 weeks
  Change in Plasma Osmolality
Blood Biomarker - Plasma Electrolyte Concentration | Through Study completion, an average of 2 weeks
  Change in Electrolyte Concentration
Blood Biomarker - Plasma Glucose Concentration | Through Study completion, an average of 2 weeks
  Change in Plasma Glucose Concentration
Body Temperature | Through Study Completion, as average of 2 weeks
  Change in degrees Celsius

OTHER OUTCOMES:
Body Composition | Through Study completion, an average of 2 weeks
  Change in Body Composition as measured by Bioimpedance Analyzer
Reaction Time | Through Study completion, an average of 2 weeks
  Change in Reaction Time
Handgrip Strength | Through Study completion, an average of 2 weeks
  Change in handgrip strength as measured by hand dynamometer
Urine Volume | Through Study completion, an average of 2 weeks
  Urine Collection
Hydration Status Saliva | Through Study completion, an average of 2 weeks
  Change in Saliva Osmolality
Heart Rate | Through Study completion, an average of 2 weeks
  Changes in heart rate as measured beats per minute
Blood Pressure | Through Study completion, an average of 2 weeks
  Change in Blood Pressure as measured systolic/diastolic mm Hg
Thirst Sensation Scale | Through Study completion, an average of 2 weeks
  Participant completed categorical scale based on "not thirsty at all" to "very, very thirsty"
Gagge Thermal Scale | Through Study completion, an average of 2 weeks
  Change in participant reported comfort (scored 1 Comfortable to 4 Very Uncomfortable) and sensation (scored 1 Cold to 7 Hot)
Urine Color | Through Study completion, an average of 2 weeks
  Participant reported color match of 8 possible categories.
Palatability | Through Study completion, an average of 2 weeks
  3 participant completed palatability questions on Likert scale scored from 1 (Dislike/Not at all) to 9 (Extremely)
Adverse Events | Through Study completion, an average of 2 weeks
  Participant Experienced Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Williams, Study Chair — Abbott Nutrition
Locations (1):
- Finlay Research, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No